CLINICAL TRIAL: NCT04651036
Title: A Randomized, Double-blind, 2-period Parallel-arm Study to Assess the Immunogenicity of 2 Subcutaneous Doses of QL0605 (6 mg) Compared to 2 Subcutaneous Doses of US Neulasta P®P (6 mg) in Healthy Male and Female Subjects
Brief Title: A Phase 1 Study to Assess the Immunogenicity of QL0605 Compared to US Neulasta in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: QL0605-OVE-002
Record Dates: First submitted 2020-11-09; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pegfilgrastim biosimilar product (Experimental): QL0605 subcutaneously at a dose of 6 mg/0.6 mL.
  Interventions: Drug: QL0605
- US Neulasta (Active Comparator): US Neulasta subcutaneously at a dose of 6 mg/0.6 mL.
  Interventions: Drug: US Neulasta

INTERVENTIONS:
Drug: QL0605 — a pegfilgrastim biosimilar to US Neulasta.
  Other Names: pegfilgrastim
  Arms: Pegfilgrastim biosimilar product
Drug: US Neulasta — US Neulasta
  Other Names: pegfilgrastim
  Arms: US Neulasta

SUMMARY:
The study was an assessor-blind, balanced, parallel, randomized, two-treatment, comparative immunogenicity study of multiple doses of subcutaneous (SC) Pegfilgrastim injection (6 mg/0.6 mL; Qilu Pharmaceutical Co., Ltd. proposed biosimilar QL0605 compared to innovator product, US-Neulasta) in healthy, adult, human subjects.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, single-dose, 2-period parallel-arm study designed to assess the immunogenicity of QL0605 and US-Neulasta.

A total of 300 healthy male and female subjects aged 18-55 years (inclusive) will be included and randomized to receive either 2 s.c. doses of QL0605 or US-NeulastaP®P in a ratio of 1:1. After the Screening Period of up to 4 weeks the subject will be randomly allocated to one of the 2 parallel treatment arms. All subjects will receive 1 s.c. injection of 6 mg QL0605 or 6 mg NeulastaP®P (US) in Treatment Period 1 and 1 s.c. injection of 6 mg QL0605 or 6 mg NeulastaP®P in Treatment Period 2. The interval between doses is ≥ 42 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give written informed consent before any assessment is performed;
2. Subjects must be a healthy male or female aged 18 to 55 years (both inclusive) at the time of informed consent;
3. Body weight ≥60 kg (males) or ≥50 kg (females) at the Screening Visit;
4. The Body Mass Index (BMI) between 18.5 to 29.9 kg/m2 (inclusive) at the Screening Visit (BMI = Body weight (kg)/[Height (m)]2);
5. Absolute neutrophil count and total leukocyte count are within the normal laboratory reference ranges; platelet count, hematocrit, and haemoglobin results are not below the lower limit of laboratory reference ranges; reticulocyte count is not above the upper limit of laboratory reference ranges; all other laboratory parameters within reference ranges or showing no clinically relevant deviations as judged by the Investigator. If the results of the laboratory parameters (other than total leukocyte count, platelet count, neutrophil count, hematocrit, reticulocyte count and hemoglobin) are outside the normal reference ranges, the subject may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate for the population under study;
6. Female subjects must either be:

   * of non-childbearing potential:

     * Postmenopausal (defined as at least 1 year without any menses) prior to the Screening Visit, and the follicle stimulating hormone levels indicative of menopause according to local laboratory reference ranges at Screening, or
     * Documented permanent surgically sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) since at least 6 weeks before the Screening Visit
   * or, if of childbearing potential:

     * Agree not to try to become pregnant during the clinical study and for 49 days after the last IMP administration and
     * Must have a negative serum pregnancy test at screening and
     * If heterosexually active, agree to consistently use 2 forms of birth control (1 of which is a highly effective method† and 1 must be a barrier method‡) from screening and throughout the study period, and for 49 days after last IMP administration. The highly effective method of contraception should be stable for at least 28 days prior to first IMP administration.

       * Highly effective forms of birth control include (i.e., less than 1% failure rate per year when used consistently and correctly):
   * Consistent and correct usage of established oral contraception (this is considered highly effective, because it is used in combination with a barrier method)
   * Injected or implanted hormonal methods of contraception
   * Established (with a failure rate < 1%) intrauterine device (IUD) or intrauterine system (IUS)
   * Bilateral tubal ligation
   * Any male partner that has undergone effective surgical sterilization, provided that the partner is the sole sexual partner of the female study participant
   * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments and complies with the preferred and usual lifestyle of the subject.

     ‡ Barrier methods of birth control include for males and females:
   * Condom without spermicidal foam/gel/film/cream/suppository or fat- or oil containing lubricant.
   * Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
7. Female subjects must agree not to breastfeed starting at the Screening Visit and throughout the clinical study period, and for 49 days after last IMP administration;
8. Female subjects must not donate ova starting at the Screening Visit and throughout the clinical study period, until the final Follow-up Visit;
9. Male subjects and their female spouse/partners who are of childbearing potential must be using 2 forms of birth control (1 of which is a highly effective method† and 1 must be a barrier method‡) starting at the Screening Visit and throughout the study period and for 49 days after the last IMP administration. A condom is required to be used also by vasectomized men to prevent delivery of the drug via seminal fluid;
10. Subjects must be non-smoker, or light smokers who smoke not more than 5 cigarettes or 1 cigar or 1 pipe per day and who agree to abstain from smoking while resident at the clinical unit.

Exclusion Criteria:

1. Known previous exposure to filgrastim, pegfilgrastim, granulocyte colony stimulating factor (G-CSF) or any analogue of these;
2. Positive test results for anti-PEG-GCSF-antibodies at the Screening Visit or based on historical data (not older than 3 months);
3. Known hypersensitivity to the study drug or any of its constituents (e.g., fructose intolerance), hypersensitivity to Escherichia coli derived proteins;
4. History of an acute severe allergic reaction (e.g., anaphylaxis; delayed hypersensitivity reaction); concurrent or history of moderate to severe allergy requiring medical treatment (including moderate seasonal allergies); concurrent or history of clinically significant latex allergy;
5. Current evidence of atopic eczema or allergic bronchial asthma;
6. History or current evidence of any clinically significant condition that might interfere with the distribution, metabolism or excretion of the any of the investigational drugs;
7. Concurrent or history of cardiac, hepatic, renal, gastrointestinal, respiratory, neurological, central nervous, mental disorders and/or hematological function disorders, which, in the judgment of the Investigator or any of the Sub-Investigators, may affect participation in this clinical study;
8. Clinically significant vital sign abnormalities or systolic blood pressure [BP] < 90 or > 139 mmHg, diastolic BP < 50 or > 89 mmHg, and/or pulse < 50 or > 90 beats per minute [bpm] at the Screening Visit (mean of triplicate measurements);
9. Subjects with abnormal 12-lead Electrocardiograms (ECGs) (QTcF >450 ms in males and 470 ms in females, signs of ischemia, sinus tachycardia [heart rate, HR >90] or sinus bradycardia [HR <50], ventricular conduct delay [QRS >120 ms] or others) which, in the judgment of the Investigator or any of the Sub-investigators, may be clinically relevant;
10. Renal impairment with estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2, based on creatinine clearance calculation by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
11. Any clinically relevant laboratory findings that, in the opinion of the Investigator, would preclude inclusion in the trial; including alanine aminotransferase (ALT), aspartate aminotransferase (AST), and bilirubin (total) > upper limit of normal (ULN). If any of these tests are out-of-range, the tests can be repeated once;
12. Previous or concurrent malignancy;
13. First degree relatives with hematological malignancy;
14. Clinically significant active infection within 4 weeks before IMP administration;
15. Any past or concurrent medical conditions that potentially increase the subject's risks or affect the evaluation of any study results, like medical history with evidence of clinically relevant pathology e.g., sickle cell disorders, spleen pathologies, hematologic malignancies or myelodysplastic disorders, and pulmonary illnesses such as Acute Respiratory Distress Syndrome, interstitial pneumonia, pulmonary edema, pulmonary infiltrates and pulmonary fibrosis;
16. Subject exhibiting spleen enlargement (as determined by ultrasound assessment) or other relevant abnormality which is, at the discretion of the Investigator, a contraindication for treatment with pegfilgrastim;
17. Presence of any clinically significant finding that, in the opinion of the Investigator, would preclude continuation in the study;
18. Participation (last dosing) in a previous clinical trial with an experimental drug within 3 months before the first administration of the IMP or five half lives of the drug, whichever is longer, prior to dosing;
19. Use of depot injectable solutions within 6 months before IMP administration. Hormonal depot injections for contraception or hormonal replacement therapy are allowed;
20. Intake of drugs and/or drugs with a long half-life within 4 weeks before IMP administration;
21. Positive test results for hepatitis B surface antigen (HbsAg), anti hepatitis B core (anti-HBc) antibodies indicative of active hepatitis, hepatitis A virus antibodies (immunoglobulin M [IgM]), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) type-1 and/or type-2 antibodies at the Screening Visit;
22. Has a history of chronic drug or alcohol abuse in the last 5 years before the date of administration of the IMP and/or positive urine drugs of abuse tests (phencyclidines, benzodiazepines, cocaine, amphetamines/ methamphetamines, cannabinoids, opiates, barbiturates, and tricyclic antidepressant drugs) and / or positive alcohol urine test at screening and admission;
23. Subjects who regularly consume large quantities of alcohol.

    * For Berlin unit: drinking > 168 g (males) and > 84 g (females) pure alcohol per week (10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 125 mL of wine [10%]) within 3 months prior to admission to the clinical unit;
    * For London unit: drinking > 21 units (males) and > 14 units (females) of alcohol per week (beer 5%, 259 ml = 10.36 g , wine 10% 100 ml = 8 g and Spirits 40% 35 ml = 11.20 g);
24. Not willing to abstain from xanthine-containing products from 24 hours prior to the Screening Visit and prior to the admission visit [Day -1] and during the in-house stay, and at all other times, to limit the consumption of caffeinated beverages or xanthine-containing products to no more than 6 units per day (1 unit = 120 mg of caffeine);
25. Plasma donation within 1 month before the Screening Visit or any blood donation / blood loss > 500 mL during the 3 months before the Screening Visit, or any planned blood donation during the time the subject is on study;
26. Use of any prescription drug (excluding hormonal contraceptives, hormone replacement therapy, and topical medications used for local treatment) or any over-the-counter drug (except ibuprofen and paracetamol) within the 2 weeks (or less than 5 x the half-life of that medication, whichever is longer) before the Baseline Visit in Period 1, which, in the judgment of the Investigator or Sub-Investigators, may affect participation in this clinical study; vitamins, minerals and nutritional supplements may be taken at the discretion of the Investigator;
27. Subjects being on a special diet or with significant weight loss from a weight reduction diet (e.g. more than approx. 5 kg within 1 month) before the Screening Visit or unwilling to maintain the same weight for the duration of the study;
28. Not willing to avoid poppy seeds and foods containing them for 72 hours prior to Screening and Day -1 visits;
29. A current (suspected or confirmed) pregnancy or currently nursing (women only);
30. Vulnerable subjects (i.e., persons under any administrative or legal supervision or persons kept in detention);
31. Subjects who are employees of Sponsor, clinical research organization (CRO) or who is the Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, other site staff or relative thereof directly involved in the conduct of the clinical study;
32. Subjects who are not able to read, speak and understand the German language (Berlin unit) or the English language (London unit);
33. Any psychological or emotional problems/disorders or resultant therapy that is likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements.
34. Subject has a positive PCR test result for SARS-CoV-2 before randomization.
35. Subject has clinical signs and symptoms consistent with COVID-19, e.g., fever, dry cough, dyspnea, sore throat, fatigue or confirmed current infection by appropriate laboratory test within the last 4 weeks prior to or at screening or on admission.
36. Subject who had severe course of COVID-19 (extracorporeal membrane oxygenation [ECMO], mechanically ventilated).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence (absolute and percentage) of ADA by treatment | 91 days
  Incidence (absolute and percentage) of anti-drug antibody by treatment

SECONDARY OUTCOMES:
AUC0-t | 91 days
  Area under the concentration-time curve (AUC) from time zero to last quantifiable concentration
AUCinf | 91 days
  Area under the concentration-time curve (AUC) from time zero to infinity
Cmax | 91 days
  Maximum serum concentration
tmax | 91 days
  time corresponding to the occurrence of Cmax
AUEC(0-Day41) | 41 days
  Area under the ANC-time curve (AUC) from time zero to day41
ANC Emax | 91 days
  Maximum ANC concentration

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Koernicke, MD, Principal Investigator — Parexel International GmbH Early Phase Clinical Unit Berlin
Locations (2):
- Parexel International GmbH Early Phase Clinical Unit Berlin, Berlin, Germany
- Parexel Early Phase Clinical Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided